CLINICAL TRIAL: NCT03102450
Title: Contraceptive Efficacy, Tolerance and Acceptability of a Benzalkonium Chloride Spermicide Cream In Women Aged Over 40 Years of Age
Acronym: BZK40+
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Laboratoire Innotech International (Industry)
Collaborators: ITEC Services (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PHX 401-14
Record Dates: First submitted 2017-03-27; First posted 2017-04-05 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Contraception

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Benzalkonium Chloride Spermicide Cream (Experimental): Pharmatex 1,2% vaginal cream (benzalkonium chloride 1,2g per 100g of vaginal cream)
  Interventions: Drug: Benzalkonium Chloride Spermicide Cream

INTERVENTIONS:
Drug: Benzalkonium Chloride Spermicide Cream — One dose of Pharmatex vaginal cream (benzalkonium chloride) must be used systematically before each intercourse, regardless of the cycle period, even during menstrual periods. In case of repeated acts of intercourse, an additional dose of cream must be used before each new act.
  Duration of treatment : 6 months (12 months optional)
  Other Names: Pharmatex 1,2% vaginal cream

SUMMARY:
In spite of many advantages of spermicides, there is no contraceptive efficacy study conducted with any spermicide in women aged over 40 years. That is why the aim of this study is to evaluate contraceptive efficacy, tolerance and acceptability of a spermicide with benzalkonium chloride (Pharmatex® cream) in women aged over 40 years.

DETAILED DESCRIPTION:
Not all contraceptive methods are appropriate for all situations, and the most appropriate method of birth control depends on the woman's overall health, her age, the frequency of her sexual activity, her sexual partners, her desire to have children in the future, and personal or family history of certain diseases.

A special interest should be paid to women aged over 40 years. Decreased fertility, increased cardiovascular risks and greater exposure to gynecological disorders during perimenopause have led to reassess the contraceptive methods in this age group. Official guidelines allow the use of any contraceptive method - including combined estrogen progestin contraceptives (COCs) - that it had been well tolerated previously.

However, more frequent contraindications during perimenopause can lead women to switch to other methods, such as the intrauterine device, the progestin-only contraception or sterilization. In this context, local contraception with spermicides represents an attractive alternative for perimenopausal women. Being totally safe, particularly metabolically, the use of spermicides in this age group is not restricted by national and international guidelines except in HIV high risk women or women with HIV clinical disease.

Furthermore, the lubricating effect of a galenic formulation of spermicides, such as cream, is particularly useful in cases of vaginal dryness, which is common in perimenopausal women. Lastly, spermicides may be used in combination with other local methods of contraception. Considering the contraindications to other contraceptives, particularly hormonal contraceptives, and the greater risks associated with these methods during perimenopause, spermicides could be an appropriate alternative for a large number of perimenopausal women.

Today, in spite of many advantages of spermicides, there is no contraceptive efficacy study conducted with any spermicide in women aged over 40 years. That is why the aim of this study is to evaluate contraceptive efficacy, tolerance and acceptability of a spermicide with benzalkonium chloride (Pharmatex® cream) in women aged over 40 years.

ELIGIBILITY:
Inclusion Criteria:

1. Women ≥ 40 years of age, fertile, having had at least one menstrual cycle in the course of the last three months
2. Women who were informed about the risks and benefits of all contraceptive methods, and for whom contraceptive methods other than spermicides were not suitable
3. Women who need a contraceptive method and who accept to use a spermicide for at least 6 months.
4. Women who have a negative pregnancy test at inclusion (the urinary pregnancy test should be performed at investigator's office then confirmed by a blood test performed in a local laboratory (quantitative beta hCG dosage)).))
5. Women who accept to comply with the requirements of the protocol including visits assessments and diary completion after each sexual intercourse
6. Women who have had a normal smear test < 3 years
7. Women affiliated to a public health insurance coverage
8. Women who have read, understood, dated and signed the informed consent form

Exclusion Criteria:

1. Women who are not able to understand a birth control method with Pharmatex® cream
2. Women who have had an unprotected sexual intercourse within 7 days before the Baseline Visit
3. Allergy or hypersensitivity to one of the components of Pharmatex® cream
4. Medical contraindication to pregnancy
5. Abnormal results of cervico-vaginal and/or vulvo-vaginal clinical examination (e.g. severe atrophic vaginitis etc.)
6. Women with history of > 2 induced abortions during lifetime (miscarriages and spontaneous abortions are not included)
7. Women with history of infectious vaginitis within the last 6 months
8. Women treated for STI within the last three months
9. HIV positive women and high-risk women for HIV
10. Breastfeeding women
11. Women participating or having participated in a clinical trial within four weeks prior to inclusion
12. Women deprived of liberty by a legal or administrative decision

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2017-12-26 (Actual); Primary Completion 2019-10-17 (Actual); Study Completion 2019-10-17 (Actual)

PRIMARY OUTCOMES:
Contraceptive Efficacy- PI over up to 12 months - typical use | up to 12 months after the inclusion
  Contraceptive efficacy of Pharmatex® cream expressed by the Pearl Index (PI) over up to 12 months of typical use. The Pearl Index is defined as the number of unintended pregnancies per 100 woman-years of a contraceptive method's use
  * Success: no fertilisation
  * Failure: unintended fertilisation (pregnancy or aborted pregnancy)

SECONDARY OUTCOMES:
Contraceptive Efficacy - PI over up to 12 months - perfect use | up to 12 months after the inclusion
  Contraceptive efficacy of Pharmatex® cream expressed by the Pearl Index (PI) over up to 12 months of perfect use
Contraceptive Efficacy - PI over up to 6 months - typical use | up to 6 months after the inclusion
  Contraceptive efficacy of Pharmatex® cream expressed by the Pearl Index (PI) at Visit 3 (M6) over up to 6 months of typical use
Contraceptive Efficacy - PI over up to 6 months - perfect use | up to 6 months after the inclusion
  Contraceptive efficacy of Pharmatex® cream expressed by the Pearl Index (PI) at Visit 3 (M6) over up to 6 months of perfect use
Contraceptive Efficacy - Pregnancy rate over up to 6 months - typical use | up to 6 months after the inclusion
  Contraceptive efficacy of Pharmatex® cream expressed by the rate of pregnancy over up to 6 months of typical use at Visit 3 (M6)
Contraceptive Efficacy - Pregnancy rate over up to 6 months - perfect use | up to 6 months after the inclusion
  Contraceptive efficacy of Pharmatex® cream expressed by the rate of pregnancy over up to 6 months of perfect use at Visit 3 (M6)
Contraceptive Efficacy - Pregnancy rate over up to 12 months - typical use | up to 12 months after the inclusion
  Contraceptive efficacy of Pharmatex® cream expressed by the rate of pregnancy over up to 12 months of typical use at Visit 4 (M12)
Contraceptive Efficacy - Pregnancy rate over up to 12 months - perfect use | up to 12 months after the inclusion
  Contraceptive efficacy of Pharmatex® cream expressed by the rate of pregnancy over up to 12 months of perfect use at Visit 4 (M12)
Number of adverse events | 6 or 12 months after the inclusion
  Number of adverse events during the study
Percentage of adverse events | 6 or 12 months after the inclusion
  Percentage of adverse events during the study
Acceptability - percentage of continuation | up to 6 or 12 months after the inclusion
  Evaluation of the acceptability of the treatment by percentage of continuation until the end of follow-up (at 6 months for all the women and at 12 months for women who have accepted to continue at visit 3 (M6))
Acceptability - adherence | up to 6 or 12 months after the inclusion
  Evaluation of the acceptability of the treatment through adherence: systematic use of benzalkonium chloride spermicide before each event of sexual intercourse recorded in the self-evaluation diary
Acceptability - ease of use (Likert scale) | up to 6 or 12 months after the inclusion
  Evaluation of the acceptability of the treatment (ease of use) evaluated through the self-evaluation diary (Likert scale) up to M6 (V3) and up to M12 (V4) for women who have continued for 12 months
Acceptability - lubricating effect (Likert scale) | up to 6 or 12 months after the inclusion
  Evaluation of the acceptability of the treatment through the lubricating effect (Likert scale) at the end of study visit: V3 (M6), or V4 (M12) or at intermediate visit in case of early withdrawal
Acceptability - global satisfaction of the woman (Likert scale) | 1, 2, 4, 6, 9, 12 months after the inclusion
  Evaluation of the global satisfaction of the treatment (Likert scale) by the woman at V2 (M2), V3 (M6) and V4 (M12) and during phone contacts PC1 (M1), PC2 (M4) and PC3 (M9)
Acceptability - global satisfaction of the investigator (Likert scale) | 2, 6, 12 months after the inclusion
  Evaluation of the global satisfaction of the treatment (Likert scale) by the investigator at V2 (M2), V3 (M6) and V4 (M12).

CONTACTS AND LOCATIONS:
Overall Officials: David Serfaty, MD, Principal Investigator — 9 rue Villersexel 75007 PARIS
Locations (15):
- France (10):
  - Cabinet Gynecologie, Carnoux-en-Provence
  - Cabinet de Gynecologie, Écully
  - Cabinet de Gynecologie, Lyon
  - Cabinet Gynecologie, Lyon
  - Cabinet de Gynecologie, Marseille
  - Cabinet de Gynecologie, Nantes
  - Cabinet Gynecologie, Neuilly-sur-Seine
  - Cabinet Gynecologie, Orléans
  - Cabinet Gynecologie, Paris
  - Cabinet Gynecologique, Strasbourg
- Russia (5):
  - Closed Joint-Stock Company "Heirs"/Nasledniki Ltd., Moscow
  - "The Pirogov Russian National Research Medical University", Moscow
  - A.I. Yevdokimov Moscow State University of Medicine and Dentistry", Moscow
  - FSBI "Scientific Center of Obstetrics, Gynecology and Perinatology n.a. V.I. Kulakov", Moscow
  - I.M. Sechenov First Moscow State Medical University", Moscow

IPD SHARING:
Plan to Share IPD: No